CLINICAL TRIAL: NCT00967018
Title: A Phase IIIb, Non-randomized, Open-label, Multi-Centre, Follow-on Safety Trial of Monthly Doses of Degarelix in Patients With Prostate Cancer
Brief Title: A Long Term Safety Study of Degarelix in Patients With Prostate Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FE200486 CS34; EudraCT No: 2008-006827-29
Record Dates: First submitted 2009-08-18; First posted 2009-08-27 (Estimated); Results first posted 2012-12-24 (Estimated); Last update posted 2013-01-03 (Estimated); Status verified 2013-01

CONDITIONS: Prostate Cancer
Keywords: Safety parameters; ECG, blood and urine samples; general health state
MeSH Terms: conditions — Prostatic Neoplasms | interventions — acetyl-2-naphthylalanyl-3-chlorophenylalanyl-1-oxohexadecyl-seryl-4-aminophenylalanyl(hydroorotyl)-4-aminophenylalanyl(carbamoyl)-leucyl-ILys-prolyl-alaninamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Degarelix (Experimental): The degarelix doses were administered into the abdominal wall every 28 days. For patients treated with goserelin in the previous trials (CS28, CS30 and CS31),a starting dose of 240 mg (40 mg/mL) degarelix was administered on Day 0 as two 3 mL subcutaneous (s.c.) injections. The subsequent maintenance of 80 mg (20 mg/mL) degarelix were administered as single 4 mL s.c. injections at 28 day intervals from day 28 to the end of the trial. For patients treated with degarelix in the previous trials, maintenance doses of 80 mg (20 mg/mL) degarelix were continued and were administered as single 4 mL s.c. injections at 28 day intervals to the end of the trial.
  Interventions: Drug: Degarelix

INTERVENTIONS:
Drug: Degarelix

SUMMARY:
Patients that completed any of the trials; CS27 (NCT00738673), CS28 (NCT00831233), CS30 (NCT00833248) or CS31 (NCT00884273) will be given the opportunity to receive monthly doses of degarelix until the drug is launched in their country. Safety parameters such as electrocardiogram (ECG), blood and urine samples and general health state will be studied. Note: patients completing the CS27 trial did not participate in the CS34 trial.

ELIGIBILITY:
Inclusion Criteria:

* Completed any of the trials; FE 200486 CS27, CS28, CS30 or CS31

Exclusion Criteria:

* Discontinued any of the trials: FE 200486 CS27, CS28, CS30 or CS31

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2009-08; Primary Completion 2011-11 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Support, Study Director — Ferring Pharmaceuticals
Locations (62):
- Belgium (2):
  - Institut Jules Bordet, Brussels
  - St. Elisabethziekenhuis, Turnhout
- France (19):
  - Hopital Jean Minjoz, Besançon
  - Institut Bergonié, Bordeaux
  - Centre Francois Baclesse, Caen
  - CHU Henri Mondor, Créteil
  - Centre Oscar Lambret, Lille
  - Centre Leon Berard, Lyon
  - Hopital de la Timone, Marseille
  - CRLC Val d' Aurelle - Oncology Radiotherapy, Montpellier
  - Hôpital Saint Louis - Radiotherapy Departement, Paris
  - Hôpital Tenon, Paris
  - Clinique Francheville, Périgueux
  - CHU La Milétrie - Oncology Radiotherapy, Poitiers
  - Clinique Saint Brieuc, Saint-Brieuc
  - Centre de Lutte Contre le Cancer Nantes-Atlantique Centre René Gauducheau, Saint-Herblain
  - Institut de Cancérologie de la Loire, Saint-Priest-en-Jarez
  - Centre Paul Strauss, Strasbourg
  - Centre de radiologie Saint Louis, Toulon
  - Clinique du Parc, Toulouse
  - IGR, Villejuif
- Italy (11):
  - Azienda Ospedaliero Universitaria Ospedali riuniti, Ancona
  - Policlinico S.Orsola Malpighi - Universita' degli Studi di Bologna, Bologna
  - Clinica Urologica 1 Universita Firenze, Florence
  - Fondazione IRCCS Istituto Nazionale Tumori, Milan
  - Fondazione IRCCS Ospedale Maggiore Policlinico Mangiagalli e Regina Elena, Milan
  - Azienda Ospedaliera Universitaria Federico II, Napoli
  - Azienda Ospedaliera Universitaria Policlinico Paolo Giaccone dell'Universita' degli Studi di Palermo, Palermo
  - Clinica Urologica - Azienda Ospedaliera di Perugia, Perugia
  - Azienda Ospedaliera S. Andrea - Universita' la Sapienza di Roma, Roma
  - S.C. Di Urologia - IRCCS Ospedale Casa Sollievo della Sofferenza, San Giovanni Rotondo
  - Azienda Ospedaliero Universitaria S. Giovanni Battista - Molinette, Torino
- Portugal (4):
  - Hospital Fernando da Fonseca, Amadora
  - Hospitais Universidade Coimbra, Coimbra
  - Centro Hospitalar Lisboa Norte, Hospital Santa Maria, Lisbon
  - Hospital S.João, Porto
- Spain (16):
  - Hospital Universitario Principe de Asturias, Alcalá de Henares-Madrid
  - Fundacion Hospital Alcorcón, Alcorcón
  - Fundación Puigvert, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitari Vall d´Hebron, Barcelona
  - Hospital de Basurto, Bilbao
  - Hospital Clinico Universitario S. Carlos, Madrid
  - Hospital Doce de Octubre, Madrid
  - Hospital universitario Ramón y Cajal, Madrid
  - Hospital Universitario Puerta de Hierro, Majadahonda
  - Hospital Manacor, Manacor
  - Hospital Universitario Central de Asturias, Oviedo
  - Hospital Santiago de Compostela, Santiago de Compostela
  - Hospital Virgen Macarena, Seville
  - Fundación IVO, Valencia
  - Hospital Xeral de Vigo, Vigo
- Sweden (6):
  - Investigational site, Gothenburg
  - SU/Sahlgrenska, Gothenburg
  - Helsingborgs Lasarett, Helsingborg
  - Universitetssjukhuset MAS, Malmo
  - Södertälje Sjukhus, Södertälje
  - Uppsala/Akademiska sjukhuset, Uppsala
- Turkey (Türkiye) (4):
  - Ankara University Faculty of Medicine - Sıhhıye, Ankara
  - Cerrahpasa Faculty of Medicine - Kocamustafapasa, Istanbul
  - Istanbul University Faculty of Medicine - ÇAPA, Istanbul
  - Marmara University Faculty of Medicine - Altunizade, Istanbul

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The patients were recruited from 16 sites in Belgium, France, Italy, Spain, Sweden and Turkey. The study was conducted between 31 August 2009 (FPFV) and 29 November 2011 (LPLV).
Period: Overall Study
Arm/Group | Degarelix
Started | 77
Completed | 56
Not Completed | 21
Not completed — Adverse Event | 2
Not completed — Physician Decision | 7
Not completed — Lost to Follow-up | 2
Not completed — Withdrawal by Subject | 1
Not completed — Miscellaneous Reasons | 9

BASELINE CHARACTERISTICS:
Arm/Group | Degarelix
Number analyzed (Participants) | 77
Age Continuous [Mean (Standard Deviation); unit: years] | 71.9 (7.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 77
Region of Enrollment [Number; unit: participants]
  France | 2
  Spain | 11
  Belgium | 2
  Turkey | 14
  Italy | 35
  Sweden | 13
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilogram per square meter] | 27.2 (4.2)
Gleason Score [Number; unit: Participants] — The Gleason score is a system of grading the aggressiveness of the prostate cancer and how fast it is likely to grow and spread. Scale is 2-10, with low numbers being the least aggressive and 10 being the most aggressive.
  Participants
    Gleason Score 2-4 | 1
    Gleason Score 5-6 | 18
    Gleason Score 7-10 | 58
Stage of Prostate Cancer [Number; unit: Participants] — Prostate cancer stage was classified according to the Tumor, Nodes, and Metastatic (TNM) scale to describe the extent of cancer. Localized refers to tumors without involvement of lymph nodes or metastasis. Advanced localized can be larger tumors that may involve the lymph nodes but no metastasis. Metastatic are more advanced cancers that are spreading beyond the original tumor. Some participants did not have their prostate cancer classified for the complete TNM scale (7 participants).
  Participants
    Localized | 36
    Locally Advanced | 19
    Metastatic | 15
    Not Classifiable | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Markedly Abnormal Values in Safety Laboratory Variables
Description: The figures present the number of participants who had markedly abnormal levels of safety laboratory variables. Only the laboratory variables that had at least one percentage of participants in either group with abnormal value are presented, more variables were included in the study.
Time Frame: Up to 22.5 months
Measure: Number; unit: Participants
Arm/Group | Degarelix
Number analyzed (Participants) | 77
Participants
  B-Haematocrit (Ratio) <=0.37 | 24
  B-Haemoglobin (g/L) <=115 | 6
  B-White blood cell count (10^9/L) <=2.8 | 2
  B-White blood cell count (10^9/L) >=16.0 | 1
  B-Red blood cell count (10^12/L) <=3.5 | 3
  B-Platelet count (10^9/L) <=75 | 1
  S-Aspartate aminotransferase (IU/L) >3xULN | 1
  S-Potassium (mmol/L) >=5.8 | 1
  S-Urea nitrogen (mmol/L) >=10.7 | 5

2. Primary Outcome: Number of Participants With Markedly Abnormal Values in Vital Signs and Body Weight
Description: This outcome measure included incidence of markedly abnormal changes in blood pressure (systolic and diastolic), pulse, and body weight. The table presents the number of participants with normal baseline and at least one post-baseline markedly abnormal value.
Time Frame: Up to 22.5 months
Measure: Number; unit: Participants
Arm/Group | Degarelix
Number analyzed (Participants) | 77
Participants
  Diastolic blood pressure <=50 and decrease >=15 | 1
  Diastolic blood pressure >=105 and increase >=15 | 1
  Systolic blood pressure <=90 and decrease >=20 | 1
  Systolic blood pressure >=180 and increase >=20 | 0
  Heart rate <=50 and decrease >=15 | 0
  Heart rate >=120 and increase >=15 | 1
  Body weight decrease of >=7 percent | 0
  Body weight increase of >=7 percent | 2

3. Other Pre Specified Outcome: Serum Levels of Prostate Specific Antigen (PSA)Over Time
Description: PSA levels were measured over time. The table below shows median levels at baseline (n=77 participants), 24 weeks (n=56), 36 weeks (n=58), 48 weeks (n=48), 72 weeks (n=9)
Time Frame: from baseline to 72 weeks
Population: The table below shows median levels at baseline (n=77 participants), 24 weeks (n=56), 36 weeks (n=58), 48 weeks (n=48), 72 weeks (n=9)
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Degarelix
Number analyzed (Participants) | 77
ng/mL
  Baseline (0 weeks) | 1.4 [0.05 to 431.3]
  Week 24 | 0.75 [0.05 to 58.5]
  Week 36 | 0.6 [0.05 to 508.8]
  Week 48 | 0.55 [0.05 to 606.5]
  Week 72 | 1.9 [0.05 to 168]

4. Other Pre Specified Outcome: Serum Levels of Testosterone Over Time
Description: Testosterone levels were measured over time. The table below shows median levels at baseline (n=77 participants), 24 weeks (n=68), 36 weeks (n=59), 48 weeks (n=54), 72 weeks (n=9)
Time Frame: from baseline to week 72
Population: The table below shows median levels at baseline (n=77 participants), 24 weeks (n=68), 36 weeks (n=59), 48 weeks (n=54), 72 weeks (n=9)
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Degarelix
Number analyzed (Participants) | 77
ng/mL
  Baseline (Week 0) | 0.05 [0.05 to 8.07]
  Week 24 | 0.05 [0.05 to 0.54]
  Week 36 | 0.05 [0.05 to 0.26]
  Week 48 | 0.08 [0.05 to 0.62]
  Week 72 | 0.12 [0.05 to 0.22]

ADVERSE EVENTS:
Time Frame: Baseline to end of treatment (maximum exposure to degarelix is approximately 25 months)
Description: Each participant's condition was monitored throughout the trial from the time of signing the informed consent until the end of the follow-up period. The investigator was to record all adverse events (AEs) in the AE log of the participant's Case Report Form.
Arm/Group | Degarelix
Serious Adverse Events (participants affected / at risk) | 5/77
Other Adverse Events (participants affected / at risk) | 30/77
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Degarelix (N=77)
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Vitreous haemorrhage (Eye disorders) | 1
Chest pain (General disorders) | 1
Gastroenteritis (Infections and infestations) | 1
Convulsion (Nervous system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Degarelix (N=77)
Haematochezia (Gastrointestinal disorders) | 2
Rectal tenesmus (Gastrointestinal disorders) | 2
Injection site inflammation (General disorders) | 7
Chills (General disorders) | 4
Injection site pain (General disorders) | 4
Chest pain (General disorders) | 2
Influenza (Infections and infestations) | 6
Gastroenteritis (Infections and infestations) | 2
Viral upper respiratory tract (Infections and infestations) | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4
Back pain (Musculoskeletal and connective tissue disorders) | 2
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Dizziness (Nervous system disorders) | 2
Syncope (Nervous system disorders) | 2
Hot flush (Vascular disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review the draft manuscript prior to publication and can request delay of publication where any contents are deemed patentable by the sponsor or confidential to the sponsor. Comments will be given within four weeks from receipt of the draft manuscript. Additional time may be required to allow Ferring to seek patent protection of the invention.